CLINICAL TRIAL: NCT01616615
Title: Aspirin for the Enhancement of Trophoblastic Invasion in Women With Abnormal Uterine Artery Doppler at 11-14 Weeks of Gestation
Acronym: ASAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Trial Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASAP; 2012-000622-22 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-06

CONDITIONS: Placental Insufficiency
MeSH Terms: conditions — Placental Insufficiency | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASPIRIN (Experimental): 150 mg milligram(s)/ day oral use
  Interventions: Drug: Aspirin
- PLACEBO (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aspirin — 150 mg/day oral use
  Arms: ASPIRIN
Drug: placebo — 1 capsule / day oral use
  Arms: PLACEBO

SUMMARY:
To establish wether a prophylactic intervention from first trimester with low-dose of aspirin improves trophoblastic invasion evaluated at third trimester in women defined as high-risk by abnormal uterine artery Doppler at first trimester

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old attending for routine ultrasound at first trimester of pregnancy between 11 and 14 weeks of gestation (Crown-to rump length 45-48mm)
* Single gestation
* Mean pulsatility index of the uterine arteries above the 95th percentile for our population

Exclusion Criteria:

* Pre-existing hypertension, renal or cardiovascular disease
* previous history of pre-eclampsia
* Pregestational diabetes
* Systemic lupus Erythematosus
* Gastric ulcer
* Acetylsalicylic acid or lactose hypersensitivity
* Bleeding disorders
* Fetal disorders (including chromosomal abnormalities)
* Administration of low molecular weight heparin
* Concomitant treatment with aspirin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Uterine artery mean pulsatility | at 28 weeks of gestation

SECONDARY OUTCOMES:
Pre-eclampsia | delivery
  pre-eclampsia defined as: diastolic blood pressure (DBP)> = 90 mmHg) or systolic (SBP)> = 140 mmHg on two separated determinations (> 4h) with proteinuria> 300 mg/24 h -Gestational age at debut of preeclampsia
Severe preeclampsia | at delivery
  Severe preeclampsia defined as: preeclampsia criteria + DBP> = 110 mmHg, proteinuria> 5g/24h, oligouria (<400 ml/24h), neurological symptoms (brain or visual), acute pulmonary edema (gasometric and radiological criteria), persistent epigastric pain, abnormal liver function (AST or Alanine aminotransferase(ALT)> 70 IU), analytical signs of hemolysis (LDH> 700 U / L) and / or thrombocytopenia (<100.000/ml).
Intrauterine Growth Retardation | at delivery
  Intrauterine Growth Retardation: birth weight below the 10th percentile of our population + pulsatility index in umbilical artery in the third trimester (on two separate occasions >48h)above the 95th percentile.
Significant neonatal morbidity | at delivery
  Significant neonatal morbidity (convulsions, intraventricular hemorrhage> grade III, periventricular leukomalacia, hypoxic-ischemic encephalopathy, abnormal electroencephalogram, necrotizing enterocolitis, acute renal failure (serum creatinine> 1.5 mg / dl) or heart failure (requiring inotropic agents
number of cesarean | at delivery
  Emergent cesarean section due to fetal wellbeing loss Birth weight
Neonatal acidosis | at delivery
  Neonatal acidosis (arterial pH <7.10 + Base excess(BE)> 12 milliequivalent (mEq) / L)
Perinatal mortality | 28 days post partum
  Perinatal mortality (> 22 weeks gestation, <28 days postpartum)
Days in the Neonatal Intensive Care Unit | 28 days post partum

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESC FIGUERAS, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (3):
- Spain (3):
  - Hospital Clinic of Barcelona, Barcelona, Barcelona
  - Institut Dexeus, Barcelona, Barcelona
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza